CLINICAL TRIAL: NCT01695265
Title: Feel Breathe, Restriction Device Ventilatory Nasal (COPD)
Acronym: BreatheCOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Jose Luis Gonzalez Montesinos, Principal Investigator, University of Cadiz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AC26392COPD
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Airflow Obstruction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercie oronasal breathing (ONB) (Experimental): Exercise protocol was walking on a treadmill for 10 minutes at a constant rate at 50% of VO2peak with oronasal breathing (ONB) (Without FeelBreathe device)
  Interventions: Other: Exercie oronasal breathing (ONB)
- Exercie nasal breathing through the FB (Experimental): Exercise protocol was walking on a treadmill for 10 minutes at a constant rate at 50% of VO2peak with nasal restriction using FeelBreathe device.
  Interventions: Device: Exercie nasal breathing through the FB

INTERVENTIONS:
Other: Exercie oronasal breathing (ONB) — 10 min at 50% of VO2 Peak achieve during a first incremental cardiopulmonary exercise test CPET using oronasal breathing (ONB)
  Arms: Exercie oronasal breathing (ONB)
Device: Exercie nasal breathing through the FB — Device: Feel Breathe, restriction device ventilatory nasal The Feel Breathe (FB) consisted of a small adhesive strip that is place across the bridge of the nose during exercise. The FB was place following procedures for placement as indicated by the manufacture's directions, while the placebo nasal, was placed over the nostrils of the subject, without interfering nasal breathing; thus, nasal airflow resistance was not increase. 10 min at 50% of VO2 Peak achieve during a first incremental cardiopulmonary exercise test CPET using FeelBreathe device (FB)
  Arms: Exercie nasal breathing through the FB

SUMMARY:
FEELBREATHE®, a nasal ventilatory restriction device, used during an exercise test in treadmill produces changes on breathing efficiency in patients with Chronic Obstructive Pulmonary Disease (COPD). 20 men with COPD with a forced expiratory volume in the first second between 30% and 70% of its predicted value were selected. Then, a maximal incremental cardiopulmonary exercise test was performed to determine ventilatory and cardiac parameters. During the second day, each participant conducted two tests with 30 min of rest between them. Exercise protocol was an identical walk on a treadmill for 10 minutes at a constant rate at 50% of VO2peak. Each test was performed randomnly in two different conditions: 1) oronasal breathing (ONB); and 2) nasal breathing through the FB.

DETAILED DESCRIPTION:
Rationale: A device called FeelBreahte (FB)® has been designed, developed and patented for inspiratory muscle training in dynamic situations.

Objetive: To examine the effects of FB on lung ventilation, gas exchange and heart rate during exercise in patients with COPD.

Methods: 20 men with COPD with a forced expiratory volume in the first second between 30% and 70% of its predicted value were selected. In the first visit to the laboratory, baseline static maximum inspiratory pressure and spirometry were performed previous to the exercise. Then, a maximal incremental cardiopulmonary exercise test was performed to determine ventilatory and cardiac parameters. During the second day, each participant conducted two tests with 30 min of rest between them. Exercise protocol was an identical walk on a treadmill for 10 minutes at a constant rate at 50% of VO2peak. Each test was performed randomnly in two different conditions: 1) oronasal breathing (ONB); and 2) nasal breathing through the FB.

Results: Lung ventilation and gas exchange during exercise in COPD patients was modified during exercise using FB. Our results showed a positive effects of FB vs ONB on dynamic hyperinflation, an improved breathing pattern and breathing efficiency, higher expiratory and inspiratory time and higher perceived effort. Despite these differences, blood oxygen saturation percentage, oxygen uptake and heart rate showed similar response between both conditions.

Conclusions: The new device FB used during exercise in COPD patients influenced ventilatory responses to an efficiency breathing compared to oronasal mode.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed of Chronic Obstructive Pulmonary Disease (COPD) at least 6 months before, with a forced expiratory volume in the first second (FEV1) between 70 and 30% of predicted value

Exclusion Criteria:

* Suffer other illness.
* Unwillingness to complete the study requirements.
* Cardiovascular diseases (resting electrocardiogram and during exercise).
* Elevated resting blood pressure (>130/85 mmHg). All inclusion and exclusion criteria were assessed by a detailed medical history and, where noted, by specific measurements.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Overall impact of a restriction device ventilatory nasal over different physiological variables in COPD | Subjects were assessed during 8 weeks
  The investigators measure minute ventilation, peak oxygen uptake (VO2p), peak carbon dioxide production (VCO2p), breathing frequency (BF), ventilatory equivalent for carbon dioxide (CO2 Eq), ventilatory equivalent for oxygen (Eq O2), expiratory tidal volume (Vtexp), inspiratory tidal volume (Vtins), end-tidal carbon dioxide tension (PETCO2), end-tidal oxygen tension (PETO2), inspiratory time (T.in), ratio of inspiratory duration to total breath duration (ti/t), expiratory time (Tex), oxygen saturation measure by pulse-oximetry SpO2), heart rate (HR), duration of the test and dyspnea and leg fatigue measures by Borg scale. Each subject performed two identical submaximal exercises at 50% of VO2peak under different breathing conditions: 1) nasal breathing with FB and 2) oronasal breathing without FB. Incremental exercise tests were performed on a treadmill ergometer using a one minute step protocol to a symptom-limited maximum.

SECONDARY OUTCOMES:
Maximal Oxygen uptake | Subjects were assessed during 8 weeks
  Before experimental trials each subject performed an incremental protocol on a treadmill ergometer (MONARK, Hamburg, Germany) for the determination of gas exchange. The test was stopped upon volitional fatigue of the subject. Gas-exchange data were measured breath by breath using an Oxycon cardiopulmonary exercise system (Jaeger, Hoechberg, Germany).
Maximum static inspiratory pressure (PImax) | Subjects were assessed during 8 weeks
  Inspiratory muscle testing was performed using a mouth pressure meter (Micro Medical Inc., Chatham, Kent, UK). The manufacturer states that the test-retest reliability of this device is ±3%. PImax was measured at residual volume and the best result from three inspiratory attempts was taken. Al least one minute was allowed between attempts to minimize the effects of muscle fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelio Arnedillo Muñoz, PhD, Study Director — Hospital Puerta del Mar Cádiz Spain; Carmen Vaz Pardal, MD, Study Director — Centro de Medicina del Deporte. Junta de Andalucía. Cádiz; Jose Lopez Chicharro, PhD, Study Director — Universidad Autonoma de Madrid; Pelayo Arroyo García, PhD, Study Chair — University of Cadiz; Jose Castro Piñero, PhD, Study Director — University of Cadiz; Jorge dR Fernández Santos, PhD Student, Study Chair — University of Cadiz; Davinia Vicente Campos, PhD, Study Chair — Universidad Complutense de Madrid; José L. González Montesinos, PhD, Principal Investigator — University of Cadiz; Julio Conde Caveda, PhD, Study Chair — University of Cadiz; Jesús G Ponce González, PhD, Study Director — University of Cadiz
Locations (1):
- Centro Andaluz Medicina del Deporte, San Fernándo, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: No
All researchers included in this study could access to the database